CLINICAL TRIAL: NCT02021019
Title: Renal Denervation to Improve Outcomes in Patients With End-stage Renal
Brief Title: Renal Denervation to Improve Outcomes in Patients With End-stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 527/13; 1052470 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2013-12-16; First posted 2013-12-27 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: End-stage Renal Disease; Hypertension
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Denervation (Experimental): Renal denervation using a catheter-based Radio-frequency approach
  Interventions: Procedure: Renal Denervation
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Procedure: Renal Denervation — Renal Denervation
  Other Names: Symplicity Renal Denervation Catheter
  Arms: Renal Denervation

SUMMARY:
Sympathetic activation is a hallmark of end-stage renal disease and adversely affects cardiovascular prognosis. Hypertension is present in the vast majority of these patients and plays a key role in the progressive deterioration of renal function and in the exceedingly high rate of cardiovascular events. Selective catheter-based renal denervation has been shown to be safe and effective in attaining improved and sustained blood pressure control in patients with resistant hypertension and normal renal function. The investigators hypothesize that catheter-based renal denervation is a safe and effective intervention to achieve sustained reduction in sympathetic nerve activity, BP and target organ damage in hypertensive End-Stage Renal Disease (ESRD) patients, which will result in improved cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease
* hypertension (BP≥140/90mmHg)

Exclusion Criteria:

* Individual has renal artery anatomy that is ineligible for treatment as assessed by the interventionalist.
* Individual has experienced a myocardial infarction, unstable angina, or a cerebrovascular accident within 3 months of the screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure change | 6 months
  Difference in the reduction of systolic office blood pressure between the renal denervation and control group at 6 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Markus P Schlaich, MD, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker IDI Heart and Diabetes Institute, Melbourne, Victoria, Australia